CLINICAL TRIAL: NCT01051063
Title: Study of GSK2130579A Tumor-Antigen-Specific Cancer Immunotherapeutic in Adult Acute Myeloid Leukemia Patients With a Suboptimal Clinical Response to Induction Chemotherapy
Brief Title: Evaluation of a New Anti-cancer Immunotherapy in Adult Acute Myeloid Leukemia Patients With a Suboptimal Clinical Response to Induction Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111727; 2008-005348-17 (EudraCT Number)
Record Dates: First submitted 2009-12-08; First posted 2010-01-18 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-06

CONDITIONS: Leukaemia, Myelocytic, Acute
Keywords: adult; WT1; ASCI; complete remission with incomplete blood count recovery; partial remission; post-induction therapy; tumor antigen; Acute Myeloid Leukemia; Immunotherapy
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

ARMS (2):
- Partial Remission Group (Experimental): Adult patients in partial remission post-induction chemotherapy, who received the GSK2130579A study product, administered sequentially, as follows: Cycle 1: 6 doses, each given at 2-week intervals; Cycle 2: 6 doses, each given at 3-week intervals; Cycle 3: 4 doses, each given at 6-week intervals; Cycle 4: 4 doses, each given at 3-month intervals, followed by 4 doses each given at 6-month intervals.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2130579A
- Complete Remission Group (Experimental): Adult patients in complete remission with incomplete blood count recovery post-induction chemotherapy, who received the GSK2130579A study product, administered sequentially, as follows: Cycle 1: 6 doses, each given at 2-week intervals; Cycle 2: 6 doses, each given at 3-week intervals; Cycle 3: 4 doses, each given at 6-week intervals; Cycle 4: 4 doses, each given at 3-month intervals, followed by 4 doses each given at 6-month intervals.
  Interventions: Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2130579A

INTERVENTIONS:
Biological: GSK Biologicals' recombinant WT1 Antigen-Specific Cancer Immunotherapeutic (ASCI) GSK2130579A — Intramuscular injection
  Other Names: WT1 ASCI

SUMMARY:
The purpose of this study is to evaluate the clinical activity and safety of a WT1 Antigen-Specific Cancer Immunotherapeutic (WT1 ASCI) as post-induction therapy in adult patients with WT1-positive AML presenting a suboptimal clinical response to induction chemotherapy. The study will also assess whether this treatment induces a specific immune response to the malignancy.

DETAILED DESCRIPTION:
At least 40 patients will be enrolled in this study, divided in two cohorts of 20 patients each. One cohort will include patients in partial remission after induction therapy and one cohort will include patients in complete remission but with incomplete blood count recovery. Patients in both cohorts will receive the same study treatment according to the same administration schedule.

This protocol summary has been updated according to the Protocol Amendment 3 (dated 10 Sept 2014).

All active follow-up visits and procedures after the concluding visit, 30 days after the last treatment administration, will be stopped In addition, no more biological samples will be collected for protocol research purposes. For each biological sample already collected in the scope of this study and not tested yet, testing will not be performed by default, except if a scientific rationale remains relevant.Blood sampling for safety monitoring as per protocol will continue.

ELIGIBILITY:
Inclusion Criteria:

* The patient has cytologically proven AML as defined by the World Health Organization (WHO) classification. The pretreatment AML karyotype should be documented.
* The leukemia is a de novo or secondary AML.
* The patient's blasts cells show expression of WT1 transcript, detected by quantitative Reverse Transcription-Polymerase Chain Reaction (qRT-PCR).The patient received the following therapy according to the Institution's standard of care.

  * For patients < 60 years old: at least two induction chemotherapy treatments.
  * For patients >= 60 years old: at least one induction chemotherapy treatment or alternative treatment.
* The first ASCI administration should be given within one year after the last chemotherapy administration. All screening procedures should be completed within seven weeks before the first ASCI administration.
* In the investigator's opinion and in compliance with the Institution Hematology Tumor Board's guidances, the patient should not be eligible for any additional chemotherapy treatment before the ASCI treatment.
* The clinical status of the patient at inclusion is one of the following:

  * Partial Remission (PR)
  * Morphologic complete remission with incomplete blood count recovery (CRi)
* Written informed consent has been obtained prior to the performance of any protocol-specific procedure.
* The patient is >= 18 years of age at the time of signature of the first informed consent form.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2.
* Adequate hepatic and renal function defined as:

  * Serum bilirubin < 1.5 times the Upper Limit of Nor-mal (ULN).
  * Serum ALT < 2.5 times the ULN.
  * Calculated creatinine clearance > 50 mL/min.
* In the view of the investigator, the patient can and will comply with the requirements of the protocol.
* If the patient is female, she must be of non-childbearing potential, i.e. have a current tubal ligation, hysterectomy, ovariectomy or be post-menopausal, or if she is of childbearing potential, then she must practice adequate contraception for 30 days prior to treatment administration, have a negative pregnancy test and continue such precautions for 2 months after completion of the treatment administration series.

Exclusion Criteria:

* The patient was diagnosed with leukemic Central Nervous System (CNS) disease (e.g. before chemotherapy) or presents neurological symptoms at baseline suggestive of a CNS involvement.
* The patient has acute promyelocytic leukemia with t(15;17) (q22;q12), (PML/RARα) or variants.
* The patient has received, or is receiving, allogeneic Stem Cell Transplantation (SCT).
* The patient has received Fludarabine, Clofarabine or Cloretazine within 12 months preceding the ASCI treat-ment.
* The patient has hypercalcemia.
* The patient is known to be HIV-positive.
* The patient has symptomatic autoimmune disease such as, but not limited to multiple sclerosis, lupus, and in-flammatory bowel disease. Patients with vitiligo are not excluded.
* The patient has a history of allergic reactions likely to be exacerbated by any component of the study investigational product.
* The patient has other concurrent severe medical prob-lems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has another metastatic cancer disease.
* The patient has a history of congestive heart failure, coronary artery disease or previous myocardial infarction.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
* The patient has received any investigational or non-registered medicinal product other than the study treat-ment within 30 days preceding the first dose of study treatment or plans to receive such a drug during the study period.
* The patient requires concomitant chronic treatment (more than 7 consecutive days) with systemic corticosteroids or any other immunosuppressive agents.
* The patient is receiving full dose subcutaneous heparins or is under anti-coagulation treatment.
* For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (3):
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Nashville, Tennessee
- France (8):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Pierre-Bénite
- Germany (11):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Complete Remission Group | Partial Remission Group
Started | 12 | 5
Completed | 2 | 1
Not Completed | 10 | 4
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Termination of the study | 5 | 0
Not completed — Moved from the study site area | 1 | 0
Not completed — Other | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Complete Remission Group | Partial Remission Group | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.3) | 64.2 (8.5) | 66.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Severe Toxicities
Description: Severe toxicities (as classified according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0) during the study treatment period defined as a study product-related or possibly study product-related:
  * Grade 4 toxicity (exception: study product-related or possibly study product-related Grade 4 fatigue - including lethargy, asthenia, and malaise - had to have a duration of at least 48 hours to be taken into account).
  * Grade 3 toxicity lasting for at least 48 hours (exceptions: myalgia, arthralgia, headache, and fever, regardless of duration).
  * Grade 2 toxicity (i.e., rash, flushing, urticaria, and dyspnea). Drug fever was not part of this definition.
  * Decrease in renal function, with a calculated creatinine clearance < 40 mL/min.
  * Grade 2 cardiac ischemia/infarction (i.e., asymptomatic and testing suggesting ischemia; stable angina).
Time Frame: During the entire study (from Month 0 to Month 49)
Population: The analysis was performed on the Total Treated population, which included all enrolled patients who had been administered at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Complete Remission Group | Partial Remission Group
Number analyzed (Participants) | 12 | 5
Participants | 1 | 0

2. Primary Outcome: Number of Patients With Best Overall Response, Defined by Either Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD)
Description: CR = having < 5% blasts in aspirate sample with marrow spicules and with a count of ≥ 200 nucleated cells, no blasts with Auer rods or persistence of extramedullary disease; different phenotype (by flow cytometry) to the pre-treatment specimen; absolute neutrophil count > 1000/mm3; platelet count ≥ 100 000/mm3 and being independent of red blood cell (RBC) transfusions.
  PR = a decrease of ≤ 50% in the % of blasts in bone marrow aspirate compared to Visit 4; being independent of RBC transfusions and the absolute neutrophil ≥ 1000/mm3 and platelet counts and ≥ 100 000/mm3.
  SD = no sufficient criteria for CR, a PR or Progressive disease (PD = Reappearance of leukemic blasts in the peripheral blood; Reappearance/development of cytologically proven extramedullary disease, Appearance of new dysplastic changes, or in a bone marrow aspirate sample (with marrow spicules and with a count of ≥200 nucleated cells) of ≥5% blasts; or, in case of early progression, a higher blast % than at Visit 4).
Time Frame: During the entire study (from Month 0 to Month 49)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Complete Remission Group | Partial Remission Group
Number analyzed (Participants) | 12 | 5
Participants
  CR | 5 | 0
  PR | 0 | 3
  SD | 6 | 1
  PD | 1 | 1

3. Secondary Outcome: Anti-WT1 Seropositivity Rate
Description: Seropositivity rate was defined as the number of patients with anti-WT1 antibody concentrations greater than or equal to (≥) 9 Enzyme-Linked Immunosorbent Assay (ELISA) units per milliliter (EU/mL).
Time Frame: At baseline (PRE), weeks (W) 5, 9, 13, 15, 21, 32, 40, 54, at months 15, 18, 21, 24, 30, 36, 42 and 49 (concluding visit), as well as follow-up visits 1 to 4
Population: The analysis was performed on the Total Treated population, which included all enrolled patients who had been administered at least one dose of the study product. For the purpose of the analysis, patients were pooled into a single group and results were tabulated for the Total Treated Group.
Measure: Count of Participants; unit: Participants
Groups:
- Total Treated Group: All adult patients (who underwent either partial or complete remission after induction chemotherapy) who received the GSK2130579A study product, administered sequentially, as follows: Cycle 1: 6 doses, each given at 2-week intervals; Cycle 2: 6 doses, each given at 3-week intervals; Cycle 3: 4 doses, each given at 6-week intervals; Cycle 4: 4 doses, each given at 3-month intervals, followed by 4 doses each given at 6-month intervals.
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
Participants
  Anti-WT1 PRE: number analyzed (Participants) | 15
  Anti-WT1 PRE | 0
  Anti-WT1 Post-dose 2, Week 5: number analyzed (Participants) | 15
  Anti-WT1 Post-dose 2, Week 5 | 1
  Anti-WT1 Post-dose 4, Week 9: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 4, Week 9 | 10
  Anti-WT1 Post-dose 6, Week 13: number analyzed (Participants) | 13
  Anti-WT1 Post-dose 6, Week 13 | 12
  Anti-WT1 Post-dose 6, Week 15: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 6, Week 15 | 12
  Anti-WT1 Post-dose 8, Week 21: number analyzed (Participants) | 10
  Anti-WT1 Post-dose 8, Week 21 | 9
  Anti-WT1 Post-dose 12, Week 32: number analyzed (Participants) | 7
  Anti-WT1 Post-dose 12, Week 32 | 6
  Anti-WT1 Post-dose 13, Week 40: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 13, Week 40 | 5
  Anti-WT1 Post-dose 16, Week 54: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 16, Week 54 | 5
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15 | 3
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18: number analyzed (Participants) | 4
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18 | 3
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21 | 3
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24 | 2
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30 | 2
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36: number analyzed (Participants) | 1
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36 | 1
  Anti-WT1 Post-dose 22, Visit 26+6 months, Month 42: number analyzed (Participants) | 1
  Anti-WT1 Post-dose 22, Visit 26+6 months, Month 42 | 1
  Anti-WT1 Last dose+30 days, Month 49: number analyzed (Participants) | 7
  Anti-WT1 Last dose+30 days, Month 49 | 5
  Anti-WT1 Post-Follow-up Visit 1: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 1 | 1
  Anti-WT1 Post-Follow-up Visit 2: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 2 | 1
  Anti-WT1 Post-Follow-up Visit 3: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 3 | 0
  Anti-WT1 Post-Follow-up Visit 4: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 4 | 0

4. Secondary Outcome: Anti-WT1 Antibody Concentrations
Description: Antibody concentrations were expressed as geometric mean concentrations, measured in ELISA units per milliliter (EU/mL).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
EU/mL
  Anti-WT1 PRE: number analyzed (Participants) | 15
  Anti-WT1 PRE | 4.5 [4.5 to 4.5]
  Anti-WT1 Post-dose 2, Week 5: number analyzed (Participants) | 15
  Anti-WT1 Post-dose 2, Week 5 | 5.4 [3.7 to 7.9]
  Anti-WT1 Post-dose 4, Week 9: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 4, Week 9 | 52.0 [18.6 to 145.4]
  Anti-WT1 Post-dose 6, Week 13: number analyzed (Participants) | 13
  Anti-WT1 Post-dose 6, Week 13 | 123.8 [50.0 to 306.5]
  Anti-WT1 Post-dose 6, Week 15: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 6, Week 15 | 138.3 [65.3 to 292.8]
  Anti-WT1 Post-dose 8, Week 21: number analyzed (Participants) | 10
  Anti-WT1 Post-dose 8, Week 21 | 105.0 [35.6 to 309.7]
  Anti-WT1 Post-dose 12, Week 32: number analyzed (Participants) | 7
  Anti-WT1 Post-dose 12, Week 32 | 136.4 [29.4 to 632.2]
  Anti-WT1 Post-dose 13, Week 40: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 13, Week 40 | 113.0 [21.1 to 603.4]
  Anti-WT1 Post-dose 16, Week 54: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 16, Week 54 | 125.3 [19.7 to 796.3]
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15 | 157.1 [34.8 to 709.5]
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18: number analyzed (Participants) | 4
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18 | 51.8 [3.5 to 774.7]
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21 | 106.6 [39.9 to 284.7]
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24 | 131.6 [0.2 to 101198.4]
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30 | 102.9 [7.8 to 1352.2]
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36: number analyzed (Participants) | 1
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36 | 122.0 [NA to NA] — Only one subject was analyzed, therefore the lower and upper limits of the 95% CI could not be computed.
  Anti-WT1 Post-dose 22, Visit 26+6 months, Month 42: number analyzed (Participants) | 1
  Anti-WT1 Post-dose 22, Visit 26+6 months, Month 42 | 115.0 [NA to NA] — Only one subject was analyzed, therefore the lower and upper limits of the 95% CI could not be computed.
  Anti-WT1 Last dose+30 days, Month 49: number analyzed (Participants) | 7
  Anti-WT1 Last dose+30 days, Month 49 | 32.2 [8.3 to 124.4]
  Anti-WT1 Post-Follow-up Visit 1: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 1 | 7.0 [0.0 to 2058.0]
  Anti-WT1 Post-Follow-up Visit 2: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 2 | 7.9 [0.0 to 10745.2]
  Anti-WT1 Post-Follow-up Visit 3: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 3 | 4.5 [NA to NA] — Only one subject was analyzed, therefore the lower and upper limits of the 95% CI could not be computed.
  Anti-WT1 Post-Follow-up Visit 4: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 4 | 4.5 [NA to NA] — Only one subject was analyzed, therefore the lower and upper limits of the 95% CI could not be computed.

5. Secondary Outcome: Anti-WT1 Antibody Response
Description: The anti-WT1 antibody response was defined as:
  For initially seronegative patients, post-vaccination antibody concentration ≥ 9 EU/mL; For initially seropositive patients, post-vaccination antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
Participants
  Anti-WT1 Post-dose 2, Week 5: number analyzed (Participants) | 15
  Anti-WT1 Post-dose 2, Week 5 | 1
  Anti-WT1 Post-dose 4, Week 9: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 4, Week 9 | 10
  Anti-WT1 Post-dose 6, Week 13: number analyzed (Participants) | 13
  Anti-WT1 Post-dose 6, Week 13 | 12
  Anti-WT1 Post-dose 6, Week 15: number analyzed (Participants) | 12
  Anti-WT1 Post-dose 6, Week 15 | 12
  Anti-WT1 Post-dose 8, Week 21: number analyzed (Participants) | 10
  Anti-WT1 Post-dose 8, Week 21 | 9
  Anti-WT1 Post-dose 12, Week 32: number analyzed (Participants) | 7
  Anti-WT1 Post-dose 12, Week 32 | 6
  Anti-WT1 Post-dose 13, Week 40: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 13, Week 40 | 5
  Anti-WT1 Post-dose 16, Week 54: number analyzed (Participants) | 6
  Anti-WT1 Post-dose 16, Week 54 | 5
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 16, Visit 19+3 months, Month 15 | 3
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18: number analyzed (Participants) | 4
  Anti-WT1 Post-dose 17, Visit 21+3 months, Month 18 | 3
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21: number analyzed (Participants) | 3
  Anti-WT1 Post-dose 18, Visit 22+3 months, Month 21 | 3
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 19, Visit 23+3 months, Month 24 | 2
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30: number analyzed (Participants) | 2
  Anti-WT1 Post-dose 20, Visit 24+6 months, Month 30 | 2
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36: number analyzed (Participants) | 1
  Anti-WT1 Post-dose 21, Visit 25+6 months, Month 36 | 1
  Anti-WT1 Post dose 22, Visit 26+6 months, Month 42: number analyzed (Participants) | 1
  Anti-WT1 Post dose 22, Visit 26+6 months, Month 42 | 1
  Anti-WT1 Last dose+30 days, Month 49: number analyzed (Participants) | 6
  Anti-WT1 Last dose+30 days, Month 49 | 5
  Anti-WT1 Post-Follow-up Visit 1: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 1 | 1
  Anti-WT1 Post-Follow-up Visit 2: number analyzed (Participants) | 2
  Anti-WT1 Post-Follow-up Visit 2 | 1
  Anti-WT1 Post-Follow-up Visit 3: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 3 | 0
  Anti-WT1 Post-Follow-up Visit 4: number analyzed (Participants) | 1
  Anti-WT1 Post-Follow-up Visit 4 | 0

6. Secondary Outcome: Number of Subjects With Any and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Related = AE assessed by the investigator as causally related to the study treatment.
Time Frame: Starting with the first administration of study treatment and ending 30 days after the last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
Participants
  Any AE(s) | 15
  Related AE(s) | 10

7. Secondary Outcome: Number of Subjects With Study Treatment Failure
Description: Study treatment failure was defined as withdrawal from investigational product because of disease progression or death. Among the characteristics evaluated were: Progression, Death in absence of Relapse, Relapse or progression or Death (Progression Free Survival event), Death [An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure; therefore it did not need to be reported as an SAE], Autopsy performed and Cause of death.
Time Frame: During the entire study (from Month 0 to Month 49)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Complete Remission Group | Partial Remission Group
Number analyzed (Participants) | 12 | 5
Participants
  Progression - yes | 6 | 5
  Progression - no | 6 | 0
  Death in absence of Relapse - yes | 0 | 0
  Death in absence of Relapse - no | 12 | 5
  Progression Free Survival event - yes | 6 | 5
  Progression Free Survival event - no | 6 | 0
  Death - yes | 4 | 2
  Death - no | 8 | 3
  Autopsy performed - yes | 0 | 0
  Autopsy performed - no | 4 | 1
  Autopsy performed - unknown | 0 | 1
  Cause of death, Disease under study (AML) | 4 | 2

8. Secondary Outcome: Number of Subjects With Any or Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related = SAE assessed by the investigator as causally related to the study treatment. An event that was part of the natural course of the disease under study (i.e., disease progression, recurrence) was captured in the study as an efficacy measure, therefore, it did not need to be reported as an SAE. Death due to progressive disease was recorded on a specific form in the CRF, but not as an SAE.
Time Frame: During the entire study (from Month 0 to Month 49)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
Participants
  Any SAE(s) | 7
  Related SAE(s) | 1

9. Secondary Outcome: Number of Patients With Abnormal Hematological and Biochemical Parameters
Description: Haematological and biochemical parameters assessed were Alanine aminotransferase, Aspartate aminotransferase, Alkaline Phosphatase, Bilirubin, Creatinine, Gamma-glutamyl transpeptidase, Hemoglobin, Hypercalcemia, Hyperkalemia, Hypernatremia, Hypoalbuminemia, Hypocalcemia, Hypokalemia, Hyponatremia, Leukocytes, Lymphopenia, Neutrophils, Platelets and Proteinuria. Parameters were assessed as per the Common Terminology Criteria for adverse events (CTCAE), where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe but not life-threatening and Grade 4 = life-threatening.
Time Frame: During the entire study (Month 0 to Month 49)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Total Treated Group
Number analyzed (Participants) | 17
Participants
  Alanine aminotransferase, Grade 0 | 8
  Alanine aminotransferase, Grade 1 | 7
  Alanine aminotransferase, Grade 2 | 2
  Alanine aminotransferase, Grade 3 | 0
  Alanine aminotransferase, Grade 4 | 0
  Alanine aminotransferase, Unknown | 0
  Aspartate aminotransferase, Grade 0 | 10
  Aspartate aminotransferase, Grade 1 | 6
  Aspartate aminotransferase, Grade 2 | 1
  Aspartate aminotransferase, Grade 3 | 0
  Aspartate aminotransferase, Grade 4 | 0
  Aspartate aminotransferase, Unknown | 0
  Alkaline Phosphatase, Grade 0 | 15
  Alkaline Phosphatase, Grade 1 | 2
  Alkaline Phosphatase, Grade 2 | 0
  Alkaline Phosphatase, Grade 3 | 0
  Alkaline Phosphatase, Grade 4 | 0
  Alkaline Phosphatase, Unknown | 0
  Bilirubin, Grade 0 | 15
  Bilirubin, Grade 1 | 1
  Bilirubin, Grade 2 | 1
  Bilirubin, Grade 3 | 0
  Bilirubin, Grade 4 | 0
  Bilirubin, Unknown | 0
  Creatinine, Grade 0 | 13
  Creatinine, Grade 1 | 3
  Creatinine, Grade 2 | 1
  Creatinine, Grade 3 | 0
  Creatinine, Grade 4 | 0
  Creatinine, Unknown | 0
  Gamma-glutamyl transpeptidase, Grade 0 | 9
  Gamma-glutamyl transpeptidase, Grade 1 | 6
  Gamma-glutamyl transpeptidase, Grade 2 | 2
  Gamma-glutamyl transpeptidase, Grade 3 | 0
  Gamma-glutamyl transpeptidase, Grade 4 | 0
  Gamma-glutamyl transpeptidase, Unknown | 0
  Hemoglobin, Grade 0 | 3
  Hemoglobin, Grade 1 | 5
  Hemoglobin, Grade 2 | 4
  Hemoglobin, Grade 3 | 3
  Hemoglobin, Grade 4 | 2
  Hemoglobin, Unknown | 0
  Hypercalcemia, Grade 0 | 14
  Hypercalcemia, Grade 1 | 3
  Hypercalcemia, Grade 2 | 0
  Hypercalcemia, Grade 3 | 0
  Hypercalcemia, Grade 4 | 0
  Hypercalcemia, Unknown | 0
  Hyperkalemia, Grade 0 | 17
  Hyperkalemia, Grade 1 | 0
  Hyperkalemia, Grade 2 | 0
  Hyperkalemia, Grade 3 | 0
  Hyperkalemia, Grade 4 | 0
  Hyperkalemia, Unknown | 0
  Hypernatremia, Grade 0 | 17
  Hypernatremia, Grade 1 | 0
  Hypernatremia, Grade 2 | 0
  Hypernatremia, Grade 3 | 0
  Hypernatremia, Grade 4 | 0
  Hypernatremia, Unknown | 0
  Hypoalbuminemia, Grade 0 | 15
  Hypoalbuminemia, Grade 1 | 1
  Hypoalbuminemia, Grade 2 | 0
  Hypoalbuminemia, Grade 3 | 1
  Hypoalbuminemia, Grade 4 | 0
  Hypoalbuminemia, Unknown | 0
  Hypocalcemia, Grade 0 | 12
  Hypocalcemia, Grade 1 | 4
  Hypocalcemia, Grade 2 | 1
  Hypocalcemia, Grade 3 | 0
  Hypocalcemia, Grade 4 | 0
  Hypocalcemia, Unknown | 0
  Hypokalemia, Grade 0 | 14
  Hypokalemia, Grade 1 | 2
  Hypokalemia, Grade 2 | 0
  Hypokalemia, Grade 3 | 1
  Hypokalemia, Grade 4 | 0
  Hypokalemia, Unknown | 0
  Hyponatremia, Grade 0 | 13
  Hyponatremia, Grade 1 | 4
  Hyponatremia, Grade 2 | 0
  Hyponatremia, Grade 3 | 0
  Hyponatremia, Grade 4 | 0
  Hyponatremia, Unknown | 0
  Leukocytes, Grade 0 | 3
  Leukocytes, Grade 1 | 3
  Leukocytes, Grade 2 | 6
  Leukocytes, Grade 3 | 4
  Leukocytes, Grade 4 | 1
  Leukocytes, Unknown | 0
  Lymphopenia, Grade 0 | 3
  Lymphopenia, Grade 1 | 4
  Lymphopenia, Grade 2 | 6
  Lymphopenia, Grade 3 | 4
  Lymphopenia, Grade 4 | 0
  Lymphopenia, Unknown | 0
  Neutrophils, Grade 0 | 5
  Neutrophils, Grade 1 | 2
  Neutrophils, Grade 2 | 3
  Neutrophils, Grade 3 | 1
  Neutrophils, Grade 4 | 6
  Neutrophils, Unknown | 0
  Platelets, Grade 0 | 0
  Platelets, Grade 1 | 5
  Platelets, Grade 2 | 1
  Platelets, Grade 3 | 5
  Platelets, Grade 4 | 6
  Platelets, Unknown | 0
  Proteinuria, Grade 0 | 12
  Proteinuria, Grade 1 | 4
  Proteinuria, Grade 2 | 0
  Proteinuria, Grade 3 | 0
  Proteinuria, Grade 4 | 0
  Proteinuria, Unknown | 1

ADVERSE EVENTS:
Time Frame: Unsolicited AEs: starting with the first administration of study treatment (Week 1) and ending 30 days after the last study treatment administration (Month 49); SAEs: During the entire study (From Month 0 to Month 49).
Description: As per protocol, safety data was performed on and tabulated for the entire population (Total Treated Group).
Arm/Group | Total Treated Group
All-Cause Mortality (participants affected / at risk) | 6/17
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Treated Group (N=17)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (3)
Vascular stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Treated Group (N=17)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (3)
Induration (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site inflammation (General disorders) | 2 (2)
Injection site pain (General disorders) | 5 (7)
Injection site reaction (General disorders) | 2 (6)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Antinuclear antibody positive (Investigations) | 1 (1)
Blood creatine increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.